CLINICAL TRIAL: NCT07305259
Title: Researching Economical Adjuvants to Cancer Therapy
Acronym: REACT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Kyle Smith, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 00005291
Record Dates: First submitted 2025-11-21; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Beta-glucan; exercise; immune system; cancer
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucan (Experimental): 375mg of beta-glucan is provided daily for 4 weeks.
  Interventions: Dietary Supplement: Beta-glucan
- Placebo (Placebo Comparator): 375mg of cellulose daily for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-glucan — 375mg of beta-glucan in the form of a ground mushroom powder. The supplement is provided in capsule form.
  Arms: Beta-glucan
Dietary Supplement: Placebo — 375mg of microcrystalline cellulose in capsule form.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if beta-glucan (a dietary fiber) improves the function of the immune system in adults. It will also tell the investigators if combining beta-glucan with single bouts of exercise provides additional benefit. The main questions it aims to answer are:

1. Does beta-glucan change the ability of immune cells to recognize cancer cells?
2. Does exercise change the type of immune cells in the blood? Researchers will compare beta-glucan to a placebo (a look-alike substance with no effect) to see if beta-glucan could improve immune function against cancer.

Participants will:

1. Take beta-glucan or a placebo daily for 4 weeks.
2. Visit the laboratory for three exercise tests.
3. Provide blood samples so researchers can study immune system cells.

DETAILED DESCRIPTION:
This investigation is a randomized, placebo-controlled trial seeking to determine the extent to which acute exercise and dietary β-glucan supplementation can augment immune responses against cancer. The investigators will mechanistically determine the receptor-ligand interactions between effector lymphocytes and target cancer cells, as well as assess multiple immunotherapies alongside the intervention (e.g., ipilimumab, pembrolizumab, monalizumab). Incorporating lifestyle medicine is well known to improve patient quality of life, and early evidence suggests it may favorably impact overall survival. It is crucial that the investigators harness the immunological potential of lifestyle interventions to broadly improve immunotherapy effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Physically fit enough to engage in maximal exercise.

Exclusion Criteria:

* BMI > 40 kg/m2
* Stage 2 hypertension (140/90 mmHg)
* Type I or II diabetes
* Autoimmune diseases
* Overt cardiovascular, respiratory, or neurological disease (e.g., previous heart attack, pacemaker, heart failure, asthma)
* Hormone replacement therapy (e.g., androgens, estrogens)
* Daily medication usage that may affect immune function (e.g., beta blockers, NSAIDs, corticosteroids, allergy medications)
* Current antibiotic use
* Heavy alcohol usage (>2 drinks per day)
* Tobacco use within the last 6 months
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Self-reported pregnancy
* Prisoners

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Cellular Cytotoxicity Assessed With Flow Cytometry | At baseline, the end of treatment at four weeks, and at eight weeks after a washout phase.
  The ability of participant peripheral blood mononuclear cells (PBMCs) to kill target cancers cells in vitro. PBMCs will be co-cultured with cancer cells for four hours, and the number of cancer cells killed over time will be quantified with flow cytometry (e.g., CD71+ labeled cancer cells with compromised cell membranes).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences and Medicine, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No